CLINICAL TRIAL: NCT05505461
Title: Efficacy and Safety of PD-1 Combined With Long-term Concurrent Neoadjuvant Chemoradiotherapy and Chemotherapy in the Treatment of Resectable Locally Advanced Esophagogastric Junction Adenocarcinoma： A Phase II Study
Brief Title: Neoadjuvant Immunotherapy and Chemoradiotherapy for Locally Advanced Esophagogastric Junction Adenocarcinoma
Acronym: NICLA
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, YE Yingjiang, Director of the department of gastrointestinal surgery, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WCWKZL-001
Record Dates: First submitted 2022-08-15; First posted 2022-08-17 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Adenocarcinoma of Esophagogastric Junction
Keywords: PD-1, neoadjuvant therapy, radiotherapy
MeSH Terms: conditions — Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — Neoadjuvant Therapy; Immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant therpy (Experimental): Neoadjuvant chemoradiation plus SOX and PD-1 antibody
  Interventions: Drug: neoadjuvant Radiation plus SOX and PD-1 antibody

INTERVENTIONS:
Drug: neoadjuvant Radiation plus SOX and PD-1 antibody — Patients will be given the perioperative treatment as below once recruited:
  First, neoradiation (5w) will be given: intensity modulated radiotherapy was given for tumors and high-risk lymphatic drainage areas. PD-1 antibody will be started concurrent the radiation for 2 cycles.
  The neochemotherapy (SOX) and PD-1 antibody will be given for 2 cycles after 1 week since radiation completed ; Patients will rest 2 weeks after the last cycle of neochemotherapy, and evaluation will be performed during this time. And D2 surgery will be performed if resectable.
  SOX and PD-1 antibody will be given q3w. Adjuvant chemotherapy: We advise starting 4 cycles of SOX regimen in 3-8w after surgery.
  Other Names: Neoadjuvant Chemoradiotherapy plus Immunotherapy

SUMMARY:
The purpose of this study was to evaluate the effect and safety of concurrent PD-1 antibody-based long-term radiotherapy followed by 2 cycles SOX with PD-1 in patients with locally advanced adenocarcinoma of esophagogastric junction.

DETAILED DESCRIPTION:
The incidence of adenocarcinoma of the esophagogastric junction (AEG) is increasing in Asian countries and Western Contries. Surgical resection is the most important treatment for AEG. However, the recurrence rate is high when surgery is performed alone. The results of CLASSIC, MAGIC, FLOT4, JCOG0501, PRODIGY, RESOLVE, CROSS trial showed that perioperative chemotherapy and pre- or postoperative chemoradiotherapy significantly increase the overall survival rate and disease free survival rate compared to surgery alone. Radiotherapy and immunotherapy can increase sensitivity to each other, and several clinical studies have also showed that PD-1 antibody may significantly prolongs the life.Thus the investigators plan to conduct this clinical trial to evaluate the effect and safety of concurrent PD-1 antibody-based long-term radiotherapy followed by 2 cycles SOX with PD-1 in patients with locally advanced adenocarcinoma of esophagogastric junction.

Subjects will receive long-term radiotherapy (5w) concurrent with PD-1 antibody for 2 cycles, then receive two cycles of SOX regimen combined PD-1 after a week's rest. Surgery will be performed 2 weeks after the last cycle of neoadjuvant treatment. Adjuvant treatment will be started 3 to 8 weeks after surgery, and SOX regimen will be given for 4 cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed adenocarcinoma of esophagogastric junction, and Her-2 negative.
2. Clinically diagnosed stage T3+orN+M0, according to CT/MRI scan.
3. No prior anti-tumor treatment, including surgery, chemotherapy, radiotherapy, and targeted therapy.
4. Eastern Cooperative Oncology Group(ECOG) performance status(PS) 0-1.
5. At least one evaluable lesion in abdominal CT/MRI according to RESIST 1.1 is required.
6. Expected survival ≥6 months.
7. Adequate organ function, Hemoglobin ≥90g/L; White blood cells ≥3.0×109/L; neutrophil count ≥1.5×109/L; Platelets ≥100×109/L; Serum creatinine (SCr) ≤ 1.5 times the upper limit of normal (ULN) or creatinine clearance rate ≥ 50ml/min (Cockcroft-Gault formula); Total bilirubin (TBIL) ≤ 1.5 times the ULN; Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) level ≤ 2.5 times the ULN; Urine protein < 2+; if urine protein ≥ 2+, 24-hour urine protein quantification shows that protein must be ≤ 1 g.
8. Normal coagulation function, no active bleeding and thrombotic diseases: International Standardized Ratio INR≤1.5×ULN; Partial thromboplastin time APTT≤1.5×ULN; Prothrombin time PT≤1.5ULN;
9. Previous use of anti-tumor Chinese medicines, proprietary Chinese medicines, and immunomodulators (such as thymosin, interleukin, etc.) must be ≥ 2 weeks from the start of the study medication;
10. Female patients should not be pregnant or breast feeding. Male should contraception.
11. Able and willing to give informed consent to participate.
12. Those who are expected to have good compliance.

Exclusion Criteria:

1. Existence of other active malignant tumors within 5 years or at the same time.
2. Already received chemotherapy, radiation therapy, targeted or immunotherapy.
3. Have any active autoimmune disease or history of autoimmune disease.
4. Patients with congenital or acquired immunodeficiency.
5. Use of immunosuppressive drugs within 14 days before the study start.
6. Administer live attenuated vaccines within 4 weeks before the study start.
7. Suffering from uncontrolled cardiac clinical symptoms or diseases, such as (1) NYHA II and above heart failure (2) unstable angina pectoris (3) myocardial infarction within 1 year (4) poorly controlled arrhythmia.
8. Patients with past and current interstitial pneumonia, pneumoconiosis, radiation pneumonia, drug-related pneumonia, etc., and severely impaired lung function.
9. Suffering from active pulmonary tuberculosis.
10. Complicated severe infection within 4 weeks before the the study start, or unexplained fever >38.5°C during the screening period/before the study start.
11. Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.

13. Allergic to any drug in this study. 14. Combined with other severe, acute and chronic diseases that may increase the risk of participating.

15.Participators who had been recruited by other clinical trial within three months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Responce (pCR) Rate | Up to 6 months
  Proportion of patients with AEG who received neoadjuvant theray with radiation plus PD-1 antibody and SOX regimen and postoperative pathological examination shows pathological complete responce

SECONDARY OUTCOMES:
R0 Resection Rate | Up to 6 months
  Proportion of patients with AEG who received surgery with pathological pathological examination proved microscopically margin-negative resection
Progression Free Survival (PFS) | Up to 3 years
  Disease Free Survival was defined as the time from the date of surgery to the date of the local recurrence, and/or distant disease, or tumor-related death.
Adverse Events | Up to 6 months
  For any adverse reactions, the researchers refer to the National Cancer Institute (NCI) standard of common toxicity (CTC)
Surgery Morbidity | 30 days and 12-months after surgery
  Surgical morbidity reported according to Clavien-Dindo classification

CONTACTS AND LOCATIONS:
Overall Officials: Yingjiang Ye, MD，PhD, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No